CLINICAL TRIAL: NCT00991705
Title: An Open-label, Two-treatment, Two-period, Two-sequence, Crossover Study to Evaluate the Effect of Atorvastatin on the Pharmacokinetics of Fimasartan in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Effect of Atorvastatin on the Pharmacokinetics of Fimasartan in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Director, Boryung Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A657-BR-CT-109
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Essential Hypertension
Keywords: Fimasartan, Atorvastatin
MeSH Terms: conditions — Essential Hypertension | interventions — Atorvastatin; fimasartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (Other): Atorvastatin (7 days) → Fimasartan + Atorvastatin (7 days)
  Interventions: Drug: Atorvastatin; Drug: Fimasartan
- Group A (Other): Fimasartan (7 days) → Fimasartan + Atorvastatin (7 days)
  Interventions: Drug: Atorvastatin; Drug: Fimasartan

INTERVENTIONS:
Drug: Atorvastatin
Drug: Fimasartan

SUMMARY:
The purpose of this study is to evaluate the effect of atorvastatin on the pharmacokinetics of fimasartan.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 45 years
* sex: male
* body weight: greater than 55 kg
* written informed consent

Exclusion Criteria:

* known allergy to Fimasartan and atorvastatin
* existing cardiac or hematological diseases
* existing hepatic and renal diseases
* existing gastrointestinal diseases
* acute or chronic diseases which could affect drug absorption or metabolism history of any serious psychological disorder
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day 3 month ago
* participation in a clinical trial during the last 2 months prior to the start of the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, Study Chair — Seoul National University Hospital

REFERENCES:
- [Derived] Shin KH, Kim TE, Kim SE, Lee MG, Song IS, Yoon SH, Cho JY, Jang IJ, Shin SG, Yu KS. The effect of the newly developed angiotensin receptor II antagonist fimasartan on the pharmacokinetics of atorvastatin in relation to OATP1B1 in healthy male volunteers. J Cardiovasc Pharmacol. 2011 Nov;58(5):492-9. doi: 10.1097/FJC.0b013e31822b9092. PMID 21765368